CLINICAL TRIAL: NCT01716676
Title: Telemedicine in Sleep Breathing Disorders: a Multicenter Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Other Study IDs: SEPAR-PII2011
Record Dates: First submitted 2012-10-29; First posted 2012-10-30 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2012-10

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

ARMS (2):
- Standard CPAP follow-up (Active Comparator)
  Interventions: Other: Standard CPAP monitoring
- Telemedicine CPAP follow-up (Experimental)
  Interventions: Other: Telemedicine CPAP monitoring (webpage and televisit)

INTERVENTIONS:
Other: Telemedicine CPAP monitoring (webpage and televisit)
  Arms: Telemedicine CPAP follow-up
Other: Standard CPAP monitoring
  Arms: Standard CPAP follow-up

SUMMARY:
In recent years medicine has been enhanced by the incorporation of technological innovations from areas as diverse as cell biology, biochemistry, genetics, biophysics and bioengineering. One of the few exceptions in this rapid process of implementing technological advances occurs in clinical medicine, where its penetration is much less effective than in other scientific and professional fields, or even in everyday life. Attempts to tackle this problem have given rise to various initiatives in the US and Europe, including Spain.

There is a surprising paucity of telemedicine systems in clinical practice, especially with respect to sleep-related breathing disorders, and most particularly obstructive sleep apnea (OSA), where protocols are urgently needed to alleviate this healthcare problem represented by its under-diagnosis and comorbidity, as well as the long waiting lists for treatment. In others words, the growing awareness of sleep disorders, especially OSA, has not been accompanied by strategic changes in the cost-effective diagnosis and/or treatment of these diseases.

CPAP therapy compliance is not always appropriate. Helping patients during the first two months usually determines compliance. Therefore, the development of strategies to support the patient during the first weeks is essential. However, this "collides" with reality, where it is difficult to properly care all patients because of congested sleep units. It is therefore necessary to implement new and imaginative control schemes especially at the beginning of the treatment. Patients' follow-up performed by telemedicine technology is an option that aims to substitute the face-to-face visits or at least reduce them considerably. In a future context, the idea is that the professional in charge of CPAP patients monitoring has on his/her agenda face-to-face visits and televisits (at distance) and information which patient will provide through online questionnaires with a certain frequency.

In this sense, this project aims to analyze whether CPAP treatment compliance of OSA patients monitored by telemedicine techniques (website and televisits) is similar to that achieved by standard monitoring but more cost-effective. The study design is a multicenter randomized trial with parallel groups and blind final evaluation after CPAP treatment following two different strategies: one through conventional monitoring in the hospital (face-to-face visiting) and another by telemedicine monitoring (non-contact visiting and website).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of OSA;
* 18-75 years;
* CPAP recommendation;
* Informed consent.

Exclusion Criteria:

* Disabling hypersomnia;
* Pregnancy;
* Psychiatric disorders;
* Previous treatment with CPAP;
* Clinical instability in the previous month;
* Inability to use information technologies (computers and web).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
CPAP compliance | 6 months
Cost-effectiveness | 6 months
Quality of life | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Isetta V, Negrin MA, Monasterio C, Masa JF, Feu N, Alvarez A, Campos-Rodriguez F, Ruiz C, Abad J, Vazquez-Polo FJ, Farre R, Galdeano M, Lloberes P, Embid C, de la Pena M, Puertas J, Dalmases M, Salord N, Corral J, Jurado B, Leon C, Egea C, Munoz A, Parra O, Cambrodi R, Martel-Escobar M, Arque M, Montserrat JM; SPANISH SLEEP NETWORK. A Bayesian cost-effectiveness analysis of a telemedicine-based strategy for the management of sleep apnoea: a multicentre randomised controlled trial. Thorax. 2015 Nov;70(11):1054-61. doi: 10.1136/thoraxjnl-2015-207032. Epub 2015 Aug 26. PMID 26310452